CLINICAL TRIAL: NCT05975957
Title: Photobiomodulation Therapy to Reduce Pain and Inflammation in Patients With Gonarthrosis: a Multicenter Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Photobiomodulation Therapy to Reduce Pain and Inflammation in Patients With Gonarthrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: TERGOS PESQUISA E ENSINO S.A (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID 369-22-ORTOP-IDOR-RJ-M-I
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis; Gonarthrosis
Keywords: photobiomodulation; gonarthrosis; analgesia
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Agnosia

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter randomized, double-blind, placebo-controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FBM (Experimental): volunteers who will receive adjuvant photobiomodulation therapy (n=119)
  Interventions: Device: Photomodulation Therapy with the Light-Aid system
- Control (Placebo Comparator): volunteers who will receive placebo treatment with inert light (n=119)
  Interventions: Device: Control

INTERVENTIONS:
Device: Photomodulation Therapy with the Light-Aid system — Patients in the intervention group (FBM) will be submitted to 10 treatment sessions (twice a week/five weeks) with the Light-Aid system (Bright Photomedicine, SP, Brazil), operated in continuous mode, with 100 LEDs of 850nm wave per tip, with application time varying from 4 to 8 minutes. Irradiation parameters will be customized based on pain intensity, skin phototype and Body Mass Index (BMI).
  Arms: FBM
Device: Control — Patients in the placebo group will undergo the same therapeutic protocol as the FBM group using a device with the same appearance as the Light-Aid System, but with inert light emission. In both groups, the treatment will be administered in contact with the skin over the knee, with the patient positioned in dorsal decubitus. The three tips of the device will be positioned horizontally over the anterior region of the knee with the central tip over the patella.
  Arms: Control

SUMMARY:
Osteoarthritis (OA) is one of the main causes of chronic pain and physical disability, which directly impacts the quality of life of patients. The prevalence of OA among adults over 60 years of age is approximately 13% in women and 10% in men. Knee OA (gonarthrosis) has as main risk factors, in addition to age, female gender and obesity. Pharmacological treatment of gonarthrosis is based on approaches to reduce symptoms and/or pain, with joint replacement (arthroplasty) being reserved for more advanced forms of the disease. In general, currently available treatments have only moderate effects and low satisfaction rates among patients. Photobiomodulation Therapy (TFBM) has been used for at least 50 years by health professionals to treat a variety of clinical conditions, especially those associated with chronic pain. TFBM is a treatment using a non-ionizing light source such as Low Intensity Laser (LBI) or Light Emitting Diodes (LED), with near-infrared wavelengths. The aim of this study is to evaluate the intensity of knee pain in the short and medium term after photobiomodulation therapy in patients with gonarthrosis. In this multicenter, randomized, placebo-controlled, double-blind clinical trial, 238 volunteers with gonarthrosis grades II and III according to the Kellgren-Lawrence classification will be recruited to be administered adjuvant treatment with TFBM. The TFBM will be performed in the knee region, twice a week, for five weeks, totaling 10 sessions. Volunteers will be allocated in the intervention group (n=119) or in the placebo group, which will be treated with 10 sessions of inert light (n=119). The hypothesis is that the photobiomodulation therapy will have a positive impact, in the short and medium term, on improving pain, functionality and quality of life of patients with symptomatic gonarthrosis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is one of the main causes of chronic pain and physical disability, which directly impacts the quality of life of patients. The prevalence of OA among adults over 60 years of age is approximately 13% in women and 10% in men. Knee OA (gonarthrosis) has as main risk factors, in addition to age, female gender and obesity. It can involve all three compartments of the knee and is clinically characterized by pain and progressive impairment of cartilage, bone, synovial membrane and ligaments. Pharmacological treatment of gonarthrosis is based on approaches to reduce symptoms and/or pain, with joint replacement (arthroplasty) being reserved for more advanced forms of the disease. In general, currently available treatments have only moderate effects and low satisfaction rates among patients. Photobiomodulation Therapy (TFBM) has been used for at least 50 years by health professionals to treat a variety of clinical conditions, especially those associated with chronic pain. TFBM is a treatment using a non-ionizing light source such as Low Intensity Laser (LBI) or Light Emitting Diodes (LED), with near-infrared wavelengths. The technique does not emit heat, is painless and non-invasive and does not have significant side effects, and can be used as an adjuvant therapy to control pain associated with gonarthrosis. The aim of this study is to evaluate the intensity of knee pain in the short and medium term after photobiomodulation therapy in patients with gonarthrosis. In this multicenter, randomized, placebo-controlled, double-blind clinical trial, 238 volunteers with gonarthrosis grades II and III according to the Kellgren-Lawrence classification will be recruited to be administered adjuvant treatment with TFBM. The TFBM will be performed in the knee region, twice a week, for five weeks, totaling 10 sessions. Volunteers will be allocated in the intervention group (n=119) or in the placebo group, which will be treated with 10 sessions of inert light (n=119). The evaluations will be made before and after TFBM or placebo and will consist of (i) measurement of pain intensity through the application of questionnaires; (ii) verify the functional mobility of the knee joint and the muscle strength of the lower limb through physical tests; (iii) evaluate the quality of life and levels of anxiety and depression through the application of questionnaires; and (iv) record the consumption of medication for analgesic purposes and the frequency of physical therapy during the trial period. The hypothesis is that the photobiomodulation therapy will have a positive impact, in the short and medium term, on improving pain, functionality and quality of life of patients with symptomatic gonarthrosis. It is also expected to observe a reduction in pain on the Visual Analog Scale of more than 20% after 10 treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged between 50 and 75 years;
* Uni or bilateral symptomatic gonarthrosis grades II or III according to the Kellgren-Lawrence classification confirmed on radiographs with weight bearing in anteroposterior, lateral and axial patella. When the disease is bilateral, the knee indicated by the patient as being the most symptomatic will be included;
* Complaint of knee pain ≥4 on the Visual Analogue Scale at the time of inclusion in the study;
* Able to walk independently, with or without walking aids;
* Cognitive ability to answer questionnaires and perform physical tests;
* Agreement to participate in the study by signing the Free and Informed Consent Form (TCLE).

Exclusion Criteria:

* Diagnosis of active malignancy except basal cell carcinoma (BCC);
* Diseases or neurological conditions that compromise the ability to perform the physical tests;
* Epilepsy;
* Skin lesions on the lower limb, close to the TFBM application site;
* Tattoos on the lower limb, close to the TFBM application site;
* Unicompartmental or total knee arthroplasty in the knee included in the study;
* History of direct trauma to the knee included in the study within the last six months;
* Active systemic inflammatory disease;
* Rheumatological diseases;
* Any previous procedure with an intra-articular approach to the knee in the last six months;
* Anticipation of adopting another form of treatment during the study period, including arthroplasty;
* Patients undergoing knee shock wave treatment in the knee included in the study;
* Absence, inability or refusal to sign the informed consent form.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change of knee pain scale by at least 20% in the FBM group assessed using the Visual Analog Scale (VAS). | 18 months
  The Visual Analogue Scale (VAS) evaluation is an instrument uses a scale of 0-10 to grade pain intensity, where 0 represents no pain and 10 the worst imaginable pain. The VAS will be applied daily until the 5th week of treatment and weekly from the sixth week to three months after treatment, through an online form sent daily to the patient via cell phone using an integrated application to the RedCap system or similar.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Vianna, Principal Investigator — Instituto D'Or de Pesquisa e Ensino
Locations (1):
- Hospital Glória D'Or, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alghadir A, Omar MT, Al-Askar AB, Al-Muteri NK. Effect of low-level laser therapy in patients with chronic knee osteoarthritis: a single-blinded randomized clinical study. Lasers Med Sci. 2014 Mar;29(2):749-55. doi: 10.1007/s10103-013-1393-3. Epub 2013 Aug 3. PMID 23912778
- [Background] Botega NJ, Bio MR, Zomignani MA, Garcia C Jr, Pereira WA. [Mood disorders among inpatients in ambulatory and validation of the anxiety and depression scale HAD]. Rev Saude Publica. 1995 Oct;29(5):355-63. doi: 10.1590/s0034-89101995000500004. Portuguese. PMID 8731275
- [Background] Chow R, Armati P, Laakso EL, Bjordal JM, Baxter GD. Inhibitory effects of laser irradiation on peripheral mammalian nerves and relevance to analgesic effects: a systematic review. Photomed Laser Surg. 2011 Jun;29(6):365-81. doi: 10.1089/pho.2010.2928. Epub 2011 Apr 1. PMID 21456946
- [Background] Brosseau L, Welch V, Wells G, Tugwell P, de Bie R, Gam A, Harman K, Shea B, Morin M. Low level laser therapy for osteoarthritis and rheumatoid arthritis: a metaanalysis. J Rheumatol. 2000 Aug;27(8):1961-9. PMID 10955339
- [Background] Fitzpatrick TB. The validity and practicality of sun-reactive skin types I through VI. Arch Dermatol. 1988 Jun;124(6):869-71. doi: 10.1001/archderm.124.6.869. No abstract available. PMID 3377516
- [Background] Fukuda VO, Fukuda TY, Guimaraes M, Shiwa S, de Lima Bdel C, Martins RA, Casarotto RA, Alfredo PP, Bjordal JM, Fucs PM. SHORT-TERM EFFICACY OF LOW-LEVEL LASER THERAPY IN PATIENTS WITH KNEE OSTEOARTHRITIS: A RANDOMIZED PLACEBO-CONTROLLED, DOUBLE-BLIND CLINICAL TRIAL. Rev Bras Ortop. 2015 Dec 6;46(5):526-33. doi: 10.1016/S2255-4971(15)30407-9. eCollection 2011 Sep-Oct. PMID 27027049
- [Background] Geurts J, Juric D, Muller M, Scharen S, Netzer C. Novel Ex Vivo Human Osteochondral Explant Model of Knee and Spine Osteoarthritis Enables Assessment of Inflammatory and Drug Treatment Responses. Int J Mol Sci. 2018 Apr 28;19(5):1314. doi: 10.3390/ijms19051314. PMID 29710775
- [Background] Goldring SR. Alterations in periarticular bone and cross talk between subchondral bone and articular cartilage in osteoarthritis. Ther Adv Musculoskelet Dis. 2012 Aug;4(4):249-58. doi: 10.1177/1759720X12437353. PMID 22859924
- [Background] de Paula Gomes CAF, Politti F, de Souza Bacelar Pereira C, da Silva ACB, Dibai-Filho AV, de Oliveira AR, Biasotto-Gonzalez DA. Exercise program combined with electrophysical modalities in subjects with knee osteoarthritis: a randomised, placebo-controlled clinical trial. BMC Musculoskelet Disord. 2020 Apr 20;21(1):258. doi: 10.1186/s12891-020-03293-3. PMID 32312265
- [Background] de Paula Gomes CAF, Dibai-Filho AV, Politti F, de Oliveira AR, de Souza Bacelar Pereira C, da Silva ACB, Biasotto-Gonzalez DA. Photobiomodulation therapy and the clinical reality in Brazil: response to the letter to the editor. BMC Musculoskelet Disord. 2021 Jan 10;22(1):59. doi: 10.1186/s12891-020-03906-x. No abstract available. PMID 33423658
- [Background] Guimaraes LS, Costa LDCM, Araujo AC, Nascimento DP, Medeiros FC, Avanzi MA, Leal-Junior ECP, Costa LOP, Tomazoni SS. Photobiomodulation therapy is not better than placebo in patients with chronic nonspecific low back pain: a randomised placebo-controlled trial. Pain. 2021 Jun 1;162(6):1612-1620. doi: 10.1097/j.pain.0000000000002189. PMID 33449509
- [Background] Hamblin MR. Mechanisms and Mitochondrial Redox Signaling in Photobiomodulation. Photochem Photobiol. 2018 Mar;94(2):199-212. doi: 10.1111/php.12864. Epub 2018 Jan 19. PMID 29164625
- [Background] GBD 2016 DALYs and HALE Collaborators. Global, regional, and national disability-adjusted life-years (DALYs) for 333 diseases and injuries and healthy life expectancy (HALE) for 195 countries and territories, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1260-1344. doi: 10.1016/S0140-6736(17)32130-X. PMID 28919118
- [Background] Hedbom E, Antonsson P, Hjerpe A, Aeschlimann D, Paulsson M, Rosa-Pimentel E, Sommarin Y, Wendel M, Oldberg A, Heinegard D. Cartilage matrix proteins. An acidic oligomeric protein (COMP) detected only in cartilage. J Biol Chem. 1992 Mar 25;267(9):6132-6. PMID 1556121
- [Background] Heidari B. Knee osteoarthritis prevalence, risk factors, pathogenesis and features: Part I. Caspian J Intern Med. 2011 Spring;2(2):205-12. PMID 24024017
- [Background] Huang YY, Chen AC, Carroll JD, Hamblin MR. Biphasic dose response in low level light therapy. Dose Response. 2009 Sep 1;7(4):358-83. doi: 10.2203/dose-response.09-027.Hamblin. PMID 20011653
- [Background] Hunter DJ, Nevitt M, Losina E, Kraus V. Biomarkers for osteoarthritis: current position and steps towards further validation. Best Pract Res Clin Rheumatol. 2014 Feb;28(1):61-71. doi: 10.1016/j.berh.2014.01.007. PMID 24792945
- [Background] Jaber K, O'Leary S, Pedler A, Sterling M, McAuliffe M. Evidence of generalised mechanical hyperalgesia in patients with advanced knee osteoarthritis undergoing total knee arthroplasty. Knee. 2018 Jun;25(3):459-465. doi: 10.1016/j.knee.2018.03.002. Epub 2018 Apr 21. PMID 29685500
- [Background] Ju C, Liu R, Zhang Y, Zhang F, Sun J, Lv XB, Zhang Z. Exosomes May Be the Potential New Direction of Research in Osteoarthritis Management. Biomed Res Int. 2019 Nov 3;2019:7695768. doi: 10.1155/2019/7695768. eCollection 2019. PMID 31781642
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Kobayashi T, Yoshihara Y, Yamada H, Fujikawa K. Procollagen IIC-peptide as a marker for assessing mechanical risk factors of knee osteoarthritis: effect of obesity and varus alignment. Ann Rheum Dis. 2000 Dec;59(12):982-4. doi: 10.1136/ard.59.12.982. PMID 11087702
- [Background] Langella LG, Casalechi HL, Tomazoni SS, Johnson DS, Albertini R, Pallotta RC, Marcos RL, de Carvalho PTC, Leal-Junior ECP. Photobiomodulation therapy (PBMT) on acute pain and inflammation in patients who underwent total hip arthroplasty-a randomized, triple-blind, placebo-controlled clinical trial. Lasers Med Sci. 2018 Dec;33(9):1933-1940. doi: 10.1007/s10103-018-2558-x. Epub 2018 Jun 16. PMID 29909435
- [Background] Lin YP, Su YH, Chin SF, Chou YC, Chia WT. Light-emitting diode photobiomodulation therapy for non-specific low back pain in working nurses: A single-center, double-blind, prospective, randomized controlled trial. Medicine (Baltimore). 2020 Aug 7;99(32):e21611. doi: 10.1097/MD.0000000000021611. PMID 32769919
- [Background] Liu Q, Niu J, Li H, Ke Y, Li R, Zhang Y, Lin J. Knee Symptomatic Osteoarthritis, Walking Disability, NSAIDs Use and All-cause Mortality: Population-based Wuchuan Osteoarthritis Study. Sci Rep. 2017 Jun 12;7(1):3309. doi: 10.1038/s41598-017-03110-3. PMID 28607349
- [Background] Loeser RF, Goldring SR, Scanzello CR, Goldring MB. Osteoarthritis: a disease of the joint as an organ. Arthritis Rheum. 2012 Jun;64(6):1697-707. doi: 10.1002/art.34453. Epub 2012 Mar 5. No abstract available. PMID 22392533
- [Background] Nazari A, Moezy A, Nejati P, Mazaherinezhad A. Efficacy of high-intensity laser therapy in comparison with conventional physiotherapy and exercise therapy on pain and function of patients with knee osteoarthritis: a randomized controlled trial with 12-week follow up. Lasers Med Sci. 2019 Apr;34(3):505-516. doi: 10.1007/s10103-018-2624-4. Epub 2018 Sep 3. PMID 30178432
- [Background] Ozdemir F, Birtane M, Kokino S. The clinical efficacy of low-power laser therapy on pain and function in cervical osteoarthritis. Clin Rheumatol. 2001;20(3):181-4. doi: 10.1007/s100670170061. PMID 11434469
- [Background] Passarella S, Karu T. Absorption of monochromatic and narrow band radiation in the visible and near IR by both mitochondrial and non-mitochondrial photoacceptors results in photobiomodulation. J Photochem Photobiol B. 2014 Nov;140:344-58. doi: 10.1016/j.jphotobiol.2014.07.021. Epub 2014 Aug 21. PMID 25226343
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558
- [Background] Roos EM, Arden NK. Strategies for the prevention of knee osteoarthritis. Nat Rev Rheumatol. 2016 Feb;12(2):92-101. doi: 10.1038/nrrheum.2015.135. Epub 2015 Oct 6. PMID 26439406
- [Background] Swagerty DL Jr, Hellinger D. Radiographic assessment of osteoarthritis. Am Fam Physician. 2001 Jul 15;64(2):279-86. PMID 11476273
- [Background] Taylor DN, Winfield T, Wynd S. Low-Level Laser Light Therapy Dosage Variables vs Treatment Efficacy of Neuromusculoskeletal Conditions: A Scoping Review. J Chiropr Med. 2020 Jun;19(2):119-127. doi: 10.1016/j.jcm.2020.06.002. Epub 2020 Aug 13. PMID 33318730
- [Background] Vassao PG, de Souza ACF, da Silveira Campos RM, Garcia LA, Tucci HT, Renno ACM. Effects of photobiomodulation and a physical exercise program on the expression of inflammatory and cartilage degradation biomarkers and functional capacity in women with knee osteoarthritis: a randomized blinded study. Adv Rheumatol. 2021 Oct 16;61(1):62. doi: 10.1186/s42358-021-00220-5. PMID 34656170
- [Background] Zhang W, Nuki G, Moskowitz RW, Abramson S, Altman RD, Arden NK, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis: part III: Changes in evidence following systematic cumulative update of research published through January 2009. Osteoarthritis Cartilage. 2010 Apr;18(4):476-99. doi: 10.1016/j.joca.2010.01.013. Epub 2010 Feb 11. PMID 20170770
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159